CLINICAL TRIAL: NCT06594042
Title: Serum Preptin Level and Its Relationship with Bone Mineral Disease in Chronic Kidney Disease Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohammed Ali, principal investigator, Assiut University
Other Study IDs: preptin chronic kidney disease
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Preptin
Keywords: chronic kidney preptin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: serum preptin — serum preptin level in chronic kidney disease

SUMMARY:
Aim of the research:To identify preptin level and relationship with bone disease in chronic kidney disease patients.

DETAILED DESCRIPTION:
Preptin is a 34-aminoacid peptide derived from the E-peptide of pro-insulin-like growth factor 2 (pro-IGF2) that is co-secreted with insulin and upregulates glucose-mediated insulin secretion. High serum preptin levels were described in conditions associated with insulin resistance, such as polycystic ovary syndrome and type 2 diabetes mellitus (T2M). Insulin and also IGF2 are known to be anabolic bone hormones .

Preptin stimulates osteoblastic proliferation and increases mineralization in a concentration-independent manner in osteoblast precursor cell , Despite being associated with insulin resistance, an increased fat mass has beneficial bone effects . While the increased mechanical loading favors bone formation, adipokines and also pancreatic and gut hormones were also proposed to mediate the relationship between fat and bone. The importance of nutritional hormones in maintaining bone mass was, thus, recognized. Insulin has anabolic bone effects, and hyperinsulinemia contributes to increased bone mineral density (BMD). Similar to insulin, insulin-like growth factor 1 (IGF1) and IGF2, preptin was recently proposed to have anabolic bone activity .

End-stage renal disease (ESRD) patients present with specific bone and mineral metabolism disturbances. Chronic kidney disease-associated mineral and bone disorder accounts for increased morbidity and mortality in those patients. Biochemical markers known thus far do not effectively predict the complex bone changes that are observed in ESRD patients .

ELIGIBILITY:
Inclusion Criteria:

* both sex groups of patients with age between 18-50 years . pre end stage renal disease and end stage renal disease patients .

Exclusion Criteria:

* type 2 diabetic patients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: study setting : dialysis unit and outpatient clinic of nephrology study subjects: the study will include 96 participants dividing into three groups of patients control group, chronic kidney disease patients .
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Serum Preptin level and its relationship with bone mineral disease in chronic kidney disease patients | baseline
  To identify preptin level and relationship with bone disease in chronic kidney disease patients.

REFERENCES:
- [Background] Kaluzna M, Pawlaczyk K, Schwermer K, Hoppe K, Yusuf Ibrahim A, Czlapka-Matyasik M, Wrotkowska E, Ziemnicka K, Oko A, Ruchala M. Is Preptin a New Bone Metabolism Parameter in Hemodialysis Patients? Life (Basel). 2021 Apr 12;11(4):341. doi: 10.3390/life11040341. PMID 33921361
- [Background] Livingstone C, Borai A. Insulin-like growth factor-II: its role in metabolic and endocrine disease. Clin Endocrinol (Oxf). 2014 Jun;80(6):773-81. doi: 10.1111/cen.12446. Epub 2014 Mar 24. PMID 24593700
- [Background] Zhang M, Xuan S, Bouxsein ML, von Stechow D, Akeno N, Faugere MC, Malluche H, Zhao G, Rosen CJ, Efstratiadis A, Clemens TL. Osteoblast-specific knockout of the insulin-like growth factor (IGF) receptor gene reveals an essential role of IGF signaling in bone matrix mineralization. J Biol Chem. 2002 Nov 15;277(46):44005-12. doi: 10.1074/jbc.M208265200. Epub 2002 Sep 4. PMID 12215457
- [Background] Naot D, Cornish J. Cytokines and Hormones That Contribute to the Positive Association between Fat and Bone. Front Endocrinol (Lausanne). 2014 May 9;5:70. doi: 10.3389/fendo.2014.00070. eCollection 2014. PMID 24847313
- [Background] Reid IR. Fat and bone. Arch Biochem Biophys. 2010 Nov 1;503(1):20-7. doi: 10.1016/j.abb.2010.06.027. Epub 2010 Jul 3. PMID 20599663
- [Background] Xiao C, Li W, Lu T, Wang J, Han J. Preptin promotes proliferation and osteogenesis of MC3T3-E1 cells by upregulating beta-catenin expression. IUBMB Life. 2019 Jul;71(7):854-862. doi: 10.1002/iub.2016. Epub 2019 Feb 6. PMID 30729647
- [Background] Ungureanu MC, Bilha SC, Hogas M, Velicescu C, Leustean L, Teodoriu LC, Preda C. Preptin: A New Bone Metabolic Parameter? Metabolites. 2023 Sep 4;13(9):991. doi: 10.3390/metabo13090991. PMID 37755271